CLINICAL TRIAL: NCT04748588
Title: Canadian Trial of the Safety and Efficacy of Investigational Therapeutics for the Treatment of Nosocomial Acquired COVID-19 Patients
Brief Title: Treatment of Nosocomial COVID-19
Acronym: CATCO-NOS
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Equipoise requirement no longer met.
Sponsor: University of Calgary (Other)
Collaborators: Sunnybrook Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REB21-0096
Record Dates: First submitted 2021-02-08; First posted 2021-02-10 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2021-01

CONDITIONS: Covid19; Nosocomial Infection; SARS-CoV2 Infection
Keywords: bamlanivimab; casirivimab; imdesimab; sotrovimab
MeSH Terms: conditions — COVID-19; Cross Infection | interventions — casirivimab; bamlanivimab; sotrovimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of care (No Intervention)
- Anti SARS-CoV-2 monoclonal antibody (Experimental): Single IV administration of an anti-SARS-CoV-2 Monoclonal antibody
  Interventions: Drug: Anti-SARS-CoV-2 mAb

INTERVENTIONS:
Drug: Anti-SARS-CoV-2 mAb — Casirivimab/imdesimab 1200mg/1200mg OR sotrovimab 500mg OR bamlanivimab 700mg IV x1.
  Casirivimab/imdesimab (REGN) and sotrovimab will be the default agents used (according to local availability) unless both unavailable AND virus strain known to be native or alpha (B.1.1.7) in which case bamlanivimab can be used.
  Other Names: casirivimab/imdesimab, bamlanivimab, sotrovimab
  Arms: Anti SARS-CoV-2 monoclonal antibody

SUMMARY:
COVID-19 is a respiratory disease caused by a novel coronavirus (SARS-CoV-2) and causes substantial morbidity and mortality. Nosocomial acquisition of SARS-CoV-2 is a frequent concern across hospital settings in Canada and is associated with substantial morbidity and mortality. This clinical trial is initially designed to evaluate the role of monoclonal antibodies against the SARS-CoV-2 spike protein, for the treatment of hospitalized patients who acquire COVID19 via nosocomial infection. New treatments, as they become available, may be integrated, with appropriate adaptation of this document. The trial was initiated with the bamlanivimab product with the options of casirivimab/imdesimab and sotrovimab added as the prevalence of bamlanivimab resistant variants of concerns increased.

It is believed that monoclonal antibody treatments are most likely to be effective early in the disease course. The ability to rapidly identify and initiate such treatments in patients with nosocomial acquisition of the infection, combined with the high mortality of 25-30% experienced by this group of patients led us to propose this trial in collaboration with the CATCO national network.

The overall objective of the study is to evaluate the safety and clinical effectiveness of anti-SARS-CoV-2 monoclonal antibody treatment relative to the control arm, in patients who develop nosocomial SARS-CoV-2 infection, on need for mechanical ventilation or death.

This study is designed as a pragmatic randomized, open-label, controlled clinical trial.

Subjects will be randomized to receive either standard-of-care (control) or the study medication on a 1:2 basis. Bamlanivimab, casirivimab/imdesimab or sotrovimab will be administered intravenously as a one-time infusion after randomization. Casirivimab/imdesimab (REGN) and sotrovimab will be the default agents based on local availability unless both are unavailable AND virus strain known to be native or alpha (B.1.1.7). Incidence of infusion-related reactions in the 24 hours post administration.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Has laboratory-confirmed SARS-CoV-2 infection as determined by PCR, or other commercial or public health assay, in any specimen prior to randomization.
* Admitted to a participating centre
* Is nosocomially acquired infection, as defined by ALL of:
* COVID19 diagnosis being made on admission day three or later;
* Admitted for a reason other than COVID19;
* Within 5 days of COVID19 diagnosis based on test collection date or initial development of symptoms, which ever was earliest.

Exclusion Criteria:

* Plan for palliation within 24 hours
* Known allergy to study medication or its components (non-medicinal ingredients)
* Ordinal scale 6 or above
* Admitted to facility for non-medical reasons including primary psychiatric diagnosis or labour and delivery.
* Pregnancy or breast feeding
* Weight less than 40kg

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2021-02-12 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Proportion of participants requiring mechanical ventilation or not surviving to hospital discharge | Length of hospitalization or 60 days

SECONDARY OUTCOMES:
In-hospital death | 60 days
Need for mechanical ventilation | 60 days
Need for new intensive care admission | 60 days
Need for new oxygen administration | 60 days

CONTACTS AND LOCATIONS:
Overall Officials: Alain Tremblay, Principal Investigator — University of Calgary; Robert Fowler, Principal Investigator — University of Toronto; Srinivas Murthy, Principal Investigator — University of British Columbia
Locations (4):
- Canada (4):
  - University of Calgary, Calgary, Alberta
  - University of Alberta, Edmonton, Alberta
  - Hôpital Montfort, Ottawa, Ontario
  - Michael Garron Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kreuzberger N, Hirsch C, Chai KL, Tomlinson E, Khosravi Z, Popp M, Neidhardt M, Piechotta V, Salomon S, Valk SJ, Monsef I, Schmaderer C, Wood EM, So-Osman C, Roberts DJ, McQuilten Z, Estcourt LJ, Skoetz N. SARS-CoV-2-neutralising monoclonal antibodies for treatment of COVID-19. Cochrane Database Syst Rev. 2021 Sep 2;9(9):CD013825. doi: 10.1002/14651858.CD013825.pub2. PMID 34473343